CLINICAL TRIAL: NCT01385059
Title: A Randomized, Phase II Study Assessing Axitinib as Pre-Surgical Therapy in Patients With High Risk Prostate Cancer
Brief Title: Axitinib Before Surgery in Treating Patients With High-Risk Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10151; NCI-2011-01105 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-06-24; First posted 2011-06-29 (Estimated); Results first posted 2023-03-07 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-02

CONDITIONS: Stage III Prostate Cancer; Stage IV Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Axitinib; Enzyme-Linked Immunosorbent Assay

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (neoadjuvant enzyme inhibitor and prostatectomy) (Experimental): Patients receive axitinib PO BID on days 1-28. Patients then undergo prostatectomy and pelvic lymph node dissection. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: axitinib; Procedure: therapeutic conventional surgery; Other: enzyme-linked immunosorbent assay; Other: laboratory biomarker analysis
- Arm II (surgery) (Active Comparator): Patients undergo prostatectomy and pelvic lymph node dissection at 5-6 weeks after biopsy confirmation of prostate cancer.
  Interventions: Procedure: therapeutic conventional surgery; Other: enzyme-linked immunosorbent assay; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: axitinib — Given PO
  Other Names: AG-013736
  Arms: Arm I (neoadjuvant enzyme inhibitor and prostatectomy)
Procedure: therapeutic conventional surgery — Undergo prostatectomy and pelvic lymph node dissection
Other: enzyme-linked immunosorbent assay — Correlative studies
  Other Names: ELISA
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This randomized phase II trial studies how well axitinib works in treating patients with high-risk prostate cancer before undergoing surgery. Axitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving axitinib before surgery may make the tumor smaller and reduce the amount of normal cells that have to be removed

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if axitinib modulates pre-metastatic niche density in patients with high-risk prostate cancer.

SECONDARY OBJECTIVES:

I. To determine if pre-metastatic niche density in regional lymph nodes (LNs) is associated with progression-free survival (PFS).

II. To determine if therapy with axitinib prolongs time to biochemical recurrence.

III. To determine if phosphorylated form of signal transducer and activator of transcription (pSTAT)3 in tumor tissue is associated with biochemical recurrence.

IV. To determine if myeloid derived suppressor cell (MDSC) recruitment in tumor tissue is associated with biochemical recurrence.

V. To determine if lysyl oxidase (LOX) expression in tumor tissue is associated with biochemical recurrence.

VI. To evaluate time to metastatic recurrence.

VII. To determine the rate of erectile dysfunction and urinary incontinence (grade >= 3 for both) in the setting of preoperative axitinib therapy.

VIII. To evaluate changes in blood-based biomarkers (pSTAT3 and selected angiogenic factors) from baseline to the time of prostatectomy.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive axitinib orally (PO) twice daily (BID) on days 1-28. Patients then undergo prostatectomy and pelvic lymph node dissection. Treatment continues in the absence of disease progression or unacceptable toxicity.

ARM II: Patients undergo prostatectomy and pelvic lymph node dissection at 5-6 weeks after biopsy confirmation of prostate cancer.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of prostate cancer
* High-risk prostate cancer as defined by 1 of the 3 following criteria:

  * Baseline prostate specific antigen (PSA) > 20
  * Clinical stage >= T3a and
  * Gleason score 8-9
* Subjects must be appropriate candidates for prostatectomy and pelvic lymph node dissection, as deemed by multidisciplinary tumor team; subjects must provide informed consent to these procedures prior to initiating study treatment
* Subjects must provide written informed consent prior to performance of study-specific procedures or assessments, and must be willing to comply with treatment and follow-up; procedures conducted as part of the subject's routine clinical management (e.g., blood count, imaging study) and obtained prior to signing of informed consent may be utilized for screening or baseline purposes provided these procedures are conducted as specified in the protocol
* Absolute neutrophil count (ANC) >= 1500 cells/mm^3
* Platelets >= 100,000 cells/mm^3
* Hemoglobin >= 9.0 g/dL
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 X upper limit of normal (ULN)
* Total bilirubin =< 1.5 X ULN
* Serum creatinine =< 1.5 X ULN or calculated creatinine clearance >= 60 mL/min
* Urinary protein < 2+ by urine analysis (UA); if UA is >= 2+ for protein then a 24-hour urine collection can be done and the patient may enter only if urinary protein is < 2 g per 24 hours
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy of >= 12 weeks
* No prior systemic therapy for prostate cancer
* No evidence of preexisting uncontrolled hypertension as documented by 2 consecutive blood pressure readings taken within 1 hour; the baseline systolic blood pressure readings must be =< 140 mm mercury (Hg), and the baseline diastolic blood pressure readings must be =< 90 mm Hg; patients whose hypertension is controlled by antihypertensive therapies are eligible
* Within 2 weeks of consent (and prior to initiating systemic therapy with axitinib if randomized to that arm), patients should visit with a radiation oncologist to discuss the option of radiation therapy (potentially with concomitant androgen deprivation therapy) for high-risk disease; if the patient has met with a radiation oncologist within 3 months of study enrollment to discuss the possibility of radiation therapy for localized prostate cancer, then this will suffice; patients do not have the right to refuse consultation; if this is the case, it must be documented by the treating physician in the medical record
* Signed and dated informed consent document indicating that the patient (or legally acceptable representative) has been informed of all pertinent aspects of the trial prior to enrollment

Exclusion Criteria:

* Prior systemic therapy for prostate cancer (including by not limited to endocrine therapy; i.e., LHRH analogues, antiandrogens, etc.)
* Evidence of metastatic disease
* Prior radiation therapy for prostate cancer
* Known history of allergic reactions to axitinib or other VEGF-TKIs
* Presence of serious or uncontrollable infection
* Major surgery <4 weeks of starting the study treatment
* Gastrointestinal abnormalities including:

  * Inability to take oral medication
  * Requirement for intravenous alimentation
  * Prior surgical procedures affecting absorption including total gastric resection
  * Treatment for active peptic ulcer disease in the past 6 months
  * Active gastrointestinal bleeding, unrelated to cancer, as evidenced by hematemesis, hematochezia or melena in the past 3 months without evidence of resolution documented by endoscopy or colonoscopy
  * Malabsorption syndromes
* Current use or anticipated need for treatment with drugs that are known potent cytochrome P450 3A4 (CYP3A4) inhibitors (ie, grapefruit juice, verapamil, ketoconazole, miconazole, itraconazole, erythromycin, telithromycin, clarithromycin, indinavir, saquinavir, ritonavir, nelfinavir, lopinavir, atazanavir, amprenavir, fosamprenavir and delavirdine)
* Current use or anticipated need for treatment with drugs that are known CYP3A4 or cytochrome P450 1A2 (CYP1A2) inducers (ie, carbamazepine, dexamethasone, felbamate, omeprazole, phenobarbital, phenytoin, amobarbital, nevirapine, primidone, rifabutin, rifampin, and St. John's wort)
* Requirement of anticoagulant therapy with oral vitamin K antagonists; therapeutic use of low molecular weight heparin is allowed
* Active seizure disorder
* A serious uncontrolled medical disorder or active infection that would impair their ability to receive study treatment
* Any of the following within the 12 months prior to study drug administration: myocardial infarction, uncontrolled angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack and 6 months for deep vein thrombosis or pulmonary embolism
* Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness
* History of a malignancy (other than prostate cancer) except those treated with curative intent for skin cancer (other than melanoma), in situ breast or in situ cervical cancer, or those treated with curative intent for any other cancer with no evidence of disease for 2 years
* Dementia or significant altered mental status that would prohibit the understanding or rendering of informed consent and compliance with the requirements of this protocol
* Other severe acute or chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the patient inappropriate for entry into this study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2011-10-28 (Actual); Primary Completion 2013-10-09 (Actual); Study Completion 2013-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sumanta Pal, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

REFERENCES:
- [Derived] Pal SK, Vuong W, Zhang W, Deng J, Liu X, Carmichael C, Ruel N, Pinnamaneni M, Twardowski P, Lau C, Yu H, Figlin RA, Agarwal N, Jones JO. Clinical and Translational Assessment of VEGFR1 as a Mediator of the Premetastatic Niche in High-Risk Localized Prostate Cancer. Mol Cancer Ther. 2015 Dec;14(12):2896-900. doi: 10.1158/1535-7163.MCT-15-0367. Epub 2015 Oct 8. PMID 26450920

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Neoadjuvant Enzyme Inhibitor and Prostatectomy) | Arm II (Surgery)
Started | 4 | 7
Completed | 4 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Neoadjuvant Enzyme Inhibitor and Prostatectomy) | Arm II (Surgery) | Total
Number analyzed (Participants) | 4 | 7 | 11
Age, Continuous [Median (Full Range); unit: years] | 67 [56 to 69] | 60 [50 to 76] | 67 [50 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 4 | 7 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 7 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 3 | 6 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 7 | 11
Clinical T stage [Count of Participants; unit: Participants] — Clinical T stage of prostate cancer was from the American Joint Committee on Cancer (AJCC) tumor, node, metastasis (TNM) system. The clinical T category is the best estimate of the extent of your disease, based on the results of the physical exam and prostate biopsy, and any imaging tests you have had. Higher numbers after T (tumor) mean the cancer is more advanced.
  Participants
    Stage T1 | 2 | 4 | 6
    Stage T2 | 2 | 3 | 5
Pathologic T Stage [Count of Participants; unit: Participants] — Pathologic T stage of prostate cancer was from the American Joint Committee on Cancer (AJCC) tumor, node, metastasis (TNM) system. Pathologic T stage is based on histopathological examination-were compared and evaluated with regard to their association with LN or distant metastasis. Higher numbers after T (tumor) mean the cancer is more advanced. And within a stage, an earlier letter means a lower stage.
  Participants
    Stage T2a/b | 0 | 1 | 1
    Stage T2c | 2 | 1 | 3
    Stage T3a/b | 2 | 5 | 7
Preoperative Gleason grade [Count of Participants; unit: Participants] — The Gleason grading system is used to help evaluate the prognosis of men with prostate cancer by the results of the prostate biopsy or surgery. The pathological scores range from 2 to 10, with higher numbers indicating greater risks and higher mortality.
  Participants
    Gleason grade < 8 | 0 | 2 | 2
    Gleason grade >= 8 | 4 | 5 | 9
Baseline PSA [Count of Participants; unit: Participants]
  Baseline PSA < 20 ng/mL | 4 | 5 | 9
  Unfavorable | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Pre-metastatic Niche Density
Description: The niche density is defined as the average number of VEGF receptor 1 (VEGFR1) clusters in 8 distinct 40X microscopic fields in the regional lymph nodes of patients. We will use a two sample student's T-test to compare the primary endpoint of pre-metastatic niche density in the patients treated with axitinib, as compared to the pre-metastatic niche density in the patients enrolled on the control arm.
Time Frame: At the time of prostatectomy
Population: Caution should be taken when drawing conclusions from these data as the target sample size needed per arm was not reached.
Measure: Median (Full Range); unit: clusters/hpf
Groups:
- Arm I (Axitinib Followed by Surgery): Patients receive Axitinib PO BID on days 1-28. Patients then undergo prostatectomy and pelvic lymph node dissection. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Axitinib: Given PO
  Therapeutic conventional surgery: Undergo prostatectomy and pelvic lymph node dissection
Arm/Group | Arm I (Axitinib Followed by Surgery) | Arm II (Surgery)
Number analyzed (Participants) | 4 | 7
clusters/hpf | 75.6 [34.3 to 79.4] | 62.5 [1 to 104.4]
Statistical Analysis 1: Comparison: Arm I (Axitinib Followed by Surgery) vs Arm II (Surgery); Test type: Other; p > 0.05, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: From the initial treatment up to 60 weeks.
Arm/Group | Arm I (Neoadjuvant Enzyme Inhibitor and Prostatectomy) | Arm II (Surgery)
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/7
Other Adverse Events (participants affected / at risk) | 3/4 | 5/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Neoadjuvant Enzyme Inhibitor and Prostatectomy) (N=4) | Arm II (Surgery) (N=7)
10002272-Anemia (Blood and lymphatic system disorders) | 2 (2) | 3 (3)
10040741-Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
10000081-Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
10016256-Fatigue (General disorders) | 0 (0) | 1 (1)
10033371-Pain (General disorders) | 0 (0) | 1 (1)
10054482-Neck edema (General disorders) | 0 (0) | 1 (1)
10020639-Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
10020647-Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
10020949-Hypocalcemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
10021005-Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
10021018-Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
10021038-Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
10003988-Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
10065780-Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
10013573-Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
10036968-Prostatic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
10061461-Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0)
10011224-Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
10020772-Hypertension (Vascular disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-18): https://cdn.clinicaltrials.gov/large-docs/59/NCT01385059/Prot_SAP_000.pdf